CLINICAL TRIAL: NCT06359483
Title: A Randomized Controlled Pilot Study on the Short-Term Impact of Meal Frequency on Bone Remodeling in Healthy Adults
Brief Title: The Impact of Meal Frequency on Bone Remodeling in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Laila Albardan, Research Assistant, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 108/2021
Record Dates: First submitted 2024-03-31; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy Adults
Keywords: Bone Remodelling; P1NP; Bone Turnover Biomarkers; Meal Frequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three Meals/Day Phase (Experimental): Participants in this arm consumed three meals daily, each providing a standardized amount of calories and macronutrients. Meals were served at specific times throughout the day, and blood samples were collected at baseline, after the last day of Phase 1, and after the last day of Phase 2. This arm aimed to investigate the impact of consuming three meals daily on bone remodeling and P1NP levels.
  Interventions: Other: Meal Frequency Manipulation
- Eight Meals/Day Phase (Experimental): Participants in this arm consumed eight meals per day, with smaller portions served more frequently throughout the day than the three-meals-per-day arm. Each meal provided a standardized amount of calories and macronutrients. Blood samples were collected at the same time points as in the three-meals-per-day arm. This arm aimed to compare the effects of consuming eight meals per day versus three meals per day on bone remodeling and P1NP levels.
  Interventions: Other: Meal Frequency Manipulation

INTERVENTIONS:
Other: Meal Frequency Manipulation — The intervention involves altering meal frequency among participants. One group consumes three standardized meals per day, while the other consumes eight smaller, more frequent meals. Meals are designed to meet nutritional needs and adhere to dietary guidelines. The aim is to assess the impact of meal frequency on bone remodeling by measuring the blood biomarker P1NP at various points during the study.

SUMMARY:
The study aimed to investigate the effect of meal frequency on bone remodeling using the marker Procollagen Type 1 N-terminal propeptide (P1NP). Thirty healthy adult males from Jordan participated in a randomized controlled intervention trial. They were randomly assigned to three or eight daily meals for three consecutive days over two phases. Blood samples were obtained at the beginning and end of each phase, and P1NP levels were analyzed. The results showed a substantial drop in P1NP levels compared to the baseline, indicating that meal frequency influences bone development. There were no significant changes between the groups eating three and eight meals per day. The study emphasizes the importance of dietary patterns in bone health and advises additional research to understand the relationship between meal frequency and bone metabolism.

DETAILED DESCRIPTION:
The study looked into how meal frequency influences bone remodeling, focusing on the Procollagen Type 1 N-terminal propeptide (P1NP) marker, which indicates bone production. Bone remodeling is a continual process in which osteoclasts break down bone tissue and osteoblasts form new bone tissue. Dietary patterns are increasingly recognized as influencing bone remodeling and general bone health, with meal frequency playing an important role in bone metabolism.

To perform the study, 30 healthy adult males aged 19 to 30 were recruited from Jordan using informational flyers. They participated in a randomized controlled intervention experiment. The participants were randomly allocated to one of two groups: one group ate three meals per day and the other ate eight meals per day. This dietary pattern was followed for three consecutive days in what was referred to as Phase 1 of the study.

Following Phase 1, there was a one-week washout phase to remove any residual effects from the previous food pattern. Following the washout period, the participants were moved to an alternate meal frequency (i.e., those who had three meals per day were now eating eight, and vice versa) for another three days, known as Phase 2.

Blood samples were collected from participants at baseline (before beginning the food intervention) and after each phase of the trial. The levels of P1NP in the blood samples were determined using an enzyme-linked immunosorbent assay (ELISA), a widely used laboratory technique for detecting and quantifying chemicals.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged between 19 and 30 years
2. Absence of medical conditions affecting bone remodeling, including:

   * Hyper/hypothyroidism
   * Diabetes
   * Cancer
   * Renal problems
   * Paget's disease
   * Cushing's disease
   * Multiple myeloma
   * Rickets
   * Osteomalacia
   * Hypogonadism
   * Osteoporosis
   * Metastatic carcinoma
   * Gaucher's disease
   * Hairy cell leukemia

Exclusion Criteria:

1. Abnormal food habits, including:

   * Night eating or frequent diet changes
   * Shift work
   * Daytime sleepers
   * Irregular sleeping patterns
2. Use of medications or supplements impacting bone remodeling, calcium homeostasis, or sleep patterns
3. History of a broken or fractured bone within the last 6 months before the study
4. Exclusively enlisting male volunteers to eliminate the potential influence of maternal hormones, such as estrogen, on bone remodeling dynamics

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
The title of the primary outcome is "Procollagen Type 1 N-terminal propeptide (P1NP) Levels." | Two phases of three consecutive days with a one-week washout period. Phase 1 involved random assignment to three or eight meals per day, followed by Phase 2 with a switch in meal frequencies. Blood samples were taken at baseline and after each phase.
  P1NP is a biomarker that reflects bone formation activity, making it a key indicator of bone remodeling processes. The primary focus of the study is to analyze changes in P1NP levels in response to alterations in meal frequency, comparing levels at baseline with those observed after different meal frequency interventions. These measurements allow researchers to assess the impact of meal frequency on bone remodeling dynamics and overall bone health.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan, Amman, Jordan